CLINICAL TRIAL: NCT02155530
Title: COmparison and Modification in Neointimal Pattern Assessed by Optical Coherence Tomography With High Versus Moderate Efficacy Statin Treatment After Drug Eluting Stent Implantation: COMPASS Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0185
Record Dates: First submitted 2014-05-26; First posted 2014-06-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High efficacy statin group (homogeneous) (Experimental): homogenous neointimal pattern at baseline OCT and randomized to atorvastatin 40 mg group
  Interventions: Drug: Atorvastatin 40mg
- Low efficacy statin group (homogeneous) (Active Comparator): homogenous neointimal pattern at baseline OCT and randomized to pravastatin 20 mg group
  Interventions: Drug: pravastatin 20 mg

INTERVENTIONS:
Drug: Atorvastatin 40mg — homogenous neointimal pattern at baseline OCT and randomized to atorvastatin 40 mg group
  Other Names: Atorvastatin 40 mg (Homogeneous)
  Arms: High efficacy statin group (homogeneous)
Drug: pravastatin 20 mg — Intervention description : homogenous neointimal pattern at baseline OCT and randomized to pravastatin 20 mg group
  Other Names: Pravastatin 20 mg (Homogeneous)
  Arms: Low efficacy statin group (homogeneous)

SUMMARY:
This study is a prospective randomized trial to evaluate and compare the quantitative and qualitative characteristics of neointimal formation between high and low efficacy statin treatment after drug eluting stent (DES) implantation, in patients with homogeneous or heterogeneous neointimal pattern accessed by Optical Coherence Tomography (OCT). The investigators postulate that high efficacy statin could have superior effect on modification of neointimal pattern, compared with lower efficacy statin. Our main hypothesis is that Atorvastatin 40mg, high efficacy statin might have superior effect on modification of neointimal pattern evaluated by serially followed OCT, compared with pravastatin 20mg in patients with DES implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 20 years old
* Patients who received OCT related to clinical needs or the end point of other study
* Patients who received DES within 1 year before OCT evaluation
* Patients with homogenous or hetero neointimal pattern by OCT
* Non-statin user and moderate or low efficacy statin user

Exclusion Criteria:

* Refuse to participate
* Contraindication to statin treatment
* Women with current or potential childbearing
* Life expectancy <1 year
* High efficacy statin user (Atorvastatin 80mg or Rosuvastatin 20mg)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of neointimal patterns assessed by 1-year followed OCT | at 1 year
  Qualitative neointimal pattern measured by OCT such as restenotic tissue structure

SECONDARY OUTCOMES:
stent coverage and neointimal thickness | at 1 year
  Change of stent coverage and neointimal thickness assessed by 1-year followed OCT
Major adverse cardiac events | at 1 year
  MACE (Major adverse cardiac events) including cardiovascular/unexpected mortality, non-fatal myocardial infarction, target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea